CLINICAL TRIAL: NCT04134299
Title: An Open-Label 12-Week Food Study to Assess the Safety, Tolerability, And Physiological Effects of An Amino Acid Food Product, AXA4010, In Subjects With Sickle Cell Disease.
Brief Title: To Assess Safety, Tolerability and Physiological Effects on Structure and Function of AXA4010 in Subjects With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AXA4010-001
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-01

CONDITIONS: To Assess the Safety and Tolerabiltiy of an Amino Acid Composition in Subjects With Sickle Cell Disease; Anemia, Sickle Cell; Sickle Cell Anemia; Sickle Cell Disorders; Sickle Cell Disease
Keywords: Amino Acid; Food Study
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AXA4010 (Experimental): AXA4010
  Interventions: Dietary Supplement: AXA4010

INTERVENTIONS:
Dietary Supplement: AXA4010 — The study will initiate with approximately eight (8) adult subjects (≥18 y/o) with SCD (Cohort 1). Each subject will receive AXA4010 twice a day (BID) for 12 weeks. Safety and tolerability will be monitored, and study procedures will be performed. Analysis of safety, tolerability and laboratory assessments at week 12 would be performed. Based on the 12-week observations from at least three subjects in Cohort 1, subsequent Cohorts 2 and 3 in Part II may be initiated.

SUMMARY:
This is an open-label study to understand the safety and tolerability of AXA4010, a novel composition of amino acids in adult and adolescent subjects with sickle cell disease over 12 weeks. The study also assesses the effects of this amino acid composition on the structure and function of the vascular system. Physiological effects on structure and function will be assessed by Magnetic Resonance Imaging (MRI) to assess blood flow in the brain and kidneys and the 6-Minute walk with pulse oximetry. Changes in blood biomarkers of inflammation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and provide written informed consent
* Male and female adolescent (ages 12 to 17 inclusive) and adult (≥ 18 years of age) subjects with a prior medically documented diagnosis of sickle cell disease (SS or β0 thalassemia)
* For Cohort 2 adult subjects only, a Screening cerebral blood flow/ velocity by transcranial doppler (TCD) should be >110 cm/sec
* Subjects must show active hemolysis at the time of screening based on each of the following parameters:

  * Lactate dehydrogenase (LDH) ≥ 2x above upper limits of normal (ULN) of the age- and gender-appropriate ranges
  * Indirect bilirubin > 2x of the age- and gender-appropriate ULN
  * Absolute reticulocyte counts > 2x of the age- and gender-appropriate ULN
* Able to ambulate (without assistance or walkers etc.) in a 6- minute walk test

Exclusion Criteria:

* Ten (10) or more Vascular-Occlusive Crisis (VOC)s that required hospital or emergency room (ER) visits within the past 12 months
* Any clinically significant changes abnormalities on the screening 12-lead ECG
* Estimated glomerular filtration rate <60mL/min/1.73m2 appropriately corrected
* Hemoglobin (Hb) ≤6.0 g/dL at Screening
* Subjects on chronic transfusion regimens, or who received a transfusion within the last 2 months prior to screening
* Experienced VOC or any other sickle crises (eg acute chest syndrome, splenic sequestration, dactylitis, stroke) within the last 2 months prior to Screening
* Current or history of significant alcohol consumption
* Other poorly controlled medical conditions as judged by the Investigator
* Known sensitivity and/or history of clinically significant food intolerance/allergies to proteins (including whey, soy, casein, amino acids, etc.)
* Unable or unwilling to adhere to contraception requirements
* Any contraindications to an MRI scan for Cohort 2 only
* Any other condition that, in the opinion of the Investigator, renders the subject at risk for compliance, compromises the well-being of the subject, or hinders study completion

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Study Product-Emergent Adverse Events [Safety and Tolerability ] | Baseline to Week 12
  Incidence of study product emergent adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Change in Lactate Dehydrogenase (LDH) | Baseline to Week 12
Change Indirect Bilirubin | Baseline to Week 12
Change Absolute Reticulocyte Count | Baseline to Week 12
Changes in Renal and Cerebral blood flow via MRI (in Adult Cohort 2 Only) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Cruz, MD, Principal Investigator — Advanced Pharma CR, LLC
Locations (4):
- United States (4):
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Primary Care research, Atlanta, Georgia
  - Newark Beth Israel Medical Center, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No